CLINICAL TRIAL: NCT00088257
Title: Maternal Fatty Acids, Child Obesity, and Asthma Immunity
Status: Completed | Type: Observational
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Matthew W. Gillman, MD, SM, Professor, Department of Population Medicine, Harvard Pilgrim Health Care
Other Study IDs: 1264; R01HL075504 (NIH)
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Mother-child pairs: Subset of mother-child pairs enrolled in Project Viva, a cohort study of pregnant women and their offspring. 411 mother-child pairs with measures of lymphocyte proliferation in their cord blood samples make up the subset for this study.

SUMMARY:
To study pre- and post-natal influences on the development of childhood asthma-related immune responses.

DETAILED DESCRIPTION:
BACKGROUND:

Since most cases of asthma occur in the first few years of life, examining its pre- and early postnatal determinants is crucial. This study focuses on determinants of the developing immune system. T helper cells are of two types. Th1 cells participate in cell-mediated immunity essential for controlling intracellular infectious agents such as bacterial and viruses. Th2 cells are essential for antibody-mediated immunity to control extracellular infectious agents. The Th2 pattern, characterized by higher levels of IgE, increased production of proinflammatory cytokines such as interleukin-4 (IL-4) or IL-13, and decreased production of interferon-gamma (IFN-gamma), predominates prenatally. If it is not balanced by a Thl pattern after birth, e.g., increased IFN-7 production, risk of asthma likely increases. Early childhood immune mechanisms associated with risk of asthma may also involve non-IgE/Th2 pathways, with increased production of IL-6 or TNF-alpha. Preliminary studies have linked asthma at various ages with reduced ratio of n-3 to n-6 polyunsaturated fatty acids, increased birth weight, and overweight. Preliminary data have also linked these dietary and weight variables to systemic production of IgE and both Th2 and non-Th2 proinflammatory cytokines. Thus allergy and inflammation may be pathways through which pre- and early postnatal dietary factors influence development of asthma. However, there are virtually no prospective human data linking maternal diet or fetal/early childhood growth with the asthma-related immune response in childhood.

The study takes advantage of the resources of Project Viva, an ongoing NIH-funded prospective cohort study of pregnant women and their offspring in eastern Massachusetts. Project Viva already includes detailed dietary data on mother and infant, maternal and cord blood samples, and data on anthropometric, social, environmental, demographic, economic, psychological, and lifestyle variables. Relevant covariates are included, such as presence and severity of atopic diseases in the parents, parental smoking, infant respiratory infections, and infant environment.

DESIGN NARRATIVE:

The study examines associations of maternal gestational n-3 and n-6 fatty acid intake, fatty acid levels in umbilical cord blood, fetal growth, and early childhood overweight with markers of allergy and inflammation at the age of 3 years. These markers include allergy-specific and total plasma IgE levels and levels of proinflammatory cytokines from antigen- and mitogen-stimulated lymphocytes. This study takes advantage of the resources of Project Viva, an ongoing NIH-funded prospective cohort study of pregnant women and their offspring. Project Viva already includes detailed dietary data on mother and infant, maternal and cord blood samples, and data on anthropometric, social, environmental, demographic, economic, psychological, and lifestyle variables. This study supports several elements not otherwise funded, including adding measurement of immune outcomes at age 3 years in a subset of 370 cohort participants. Given the existing infrastructure of Project Viva, the study provides a relatively economical way to address scientific questions of major public health importance.

ELIGIBILITY:
Women were eligible for participation in Project Viva if they:

1. Were <22 weeks pregnant
2. Planned to receive prenatal care at one of the selected clinics
3. Planned to deliver at one of the two study hospitals
4. Were able to answer questions in English

Women were ineligible if they:

1. Planned to terminate their pregnancy
2. Planned to move from the local area before the end of the follow-up period
3. Were pregnant with multiples (twins, triplets, etc)

Project Viva mother-child pairs were eligible for this study if they had provided maternal dietary date during pregnancy and a cord blood sample at delivery on which lymphocyte proliferation had been measured.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women were recruited in 1999-2002 following their initial prenatal visit at one of eight obstetric offices of a multi-specialty group practice in eastern MA.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2004-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Markers of allergy and inflammation at age 3 years | Age 3 years
  Allergy-specific and total plasma IgE levels; asthma-related pro-inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gillman, Principal Investigator — Harvard Pilgrim Health Care